CLINICAL TRIAL: NCT01520285
Title: A Multi-center, Randomized, Open-label, Parallel-group Clinical Study to Compare the Effects of Lercanidipine Hydrochloride Tablet (Zanidip®) and Felodipine Sustained-Release Tablet for the Treatment of Patients With Mild-to-Moderate Hypertension
Brief Title: Compare the Effects of Lercanidipine Hydrochloride Tablet (Zanidip®) and Felodipine Sustained-Release Tablet for Hypertension
Acronym: Zanidip
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lee's Pharmaceutical Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LEES_Zanidip_1
Record Dates: First submitted 2012-01-13; First posted 2012-01-27 (Estimated); Last update posted 2014-10-16 (Estimated); Status verified 2014-10

CONDITIONS: Hypertension
Keywords: hypertension; Blood pressure decrease; efficacy
MeSH Terms: conditions — Hypertension | interventions — lercanidipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Zanidip (Active Comparator): tablets
  Interventions: Drug: Zanidip
- Control Drug (Placebo Comparator): Felodipine sustained-release tablet (5mg/tablet)
  Interventions: Drug: Felodipine sustained-release tablet

INTERVENTIONS:
Drug: Zanidip — Lercanidipine hydrochloride (10mg/tablet)once per day
  Arms: Zanidip
Drug: Felodipine sustained-release tablet — Felodipine sustained-release tablet (5mg/tablet)
  Arms: Control Drug

SUMMARY:
This study will be compare Felodipine sustained-release tablets, to Lercanidipine hydrochloride tablets (Zanidip®) for the treatment of patients with mild-to-moderate primary hypertension and to investigate the influence on patients' heart rate and blood pressure variability.

DETAILED DESCRIPTION:
The study is designed as a multicenter, randomized, open-label, parallel-group and active controlled clinical study. The ratio of test group (lercanidipine group) and control group (felodipine group) is 1:1.

The study period lasts for 8 weeks, including 0-2 weeks of run-in period and 6 weeks of treatment period. There are 5 visits: run-in period (V1), baseline (V2), 2 weeks after treatment (V3), 4 weeks after treatment (V4) and 6 weeks after treatment (V5).

There are about 2 weeks for run-in period, the patients should start continuous recording the data of self-measuring blood pressure and heart rate for 1 week (at least 5days) before randomized in V2. Patients who under the antihypertensive treatment or have discontinued the antihypertensive treatment for less than 1 week need to discontinued the treatment for over 1week and start this trial; patients who never received any antihypertensive drug or patients who have discontinued the antihypertensive treatment for over one week will directly enter treatment period.

In V2, investigator should confirm the patient meet the inclusion/exclusion criteria, only the eligible patients will be divided groups by random, and the rest need to drop-out this trial. In that day of randomization, patients should take drug.

After the randomization, the patients will be given study drugs, and take take once-daily dose of the study drugs at 07:00-09:00 (except the day of visit). During the treatment, there will be a visit every 2 weeks, and in each visit the patients need to get the study drug for next two weeks, totally 3 times. In V3 and V4, if the patients' mean DBP ≥ 90 mm Hg, the doses will be doubled, twice a day (07:00- 09:00 in the morning and 16:00-18:00 in the afternoon), otherwise, the dosage do not change.

From the day beginning administration of the study drugs, patient should measure the BP and HR every day with the electronic sphygmomanometer after getting up in the morning and before going to bed. And patient records the data of blood pressure and heart rate in the record card. 2 to 3 minutes waiting for each measure and at least 12 significant date for consecutive 3 days. In every visit, investigator will collect the data of patient's self-measuring blood pressure, and give new recording forms for self-measuring blood pressure to the patients.

ELIGIBILITY:
Inclusion Criteria:

Study population is patients with mild-to-moderate primary hypertension. The diagnosis of the patients should be in accordance with the diagnostic criteria in Chinese Guidelines for Hypertension Prevention and Treatment (2010). Patients meeting all of the following criteria are enrolled in the study:

1. Male or female patient, aged 18-75 years;
2. Mild-to-moderate primary hypertension;
3. 90mmHg ≤ DBP < 110 mmHg and SBP < 180mmHg;
4. Patient's 24h mean blood pressure (measuring by ABPM)> 130/80mmHg;
5. Patient has signed informed consent form;

Exclusion Criteria:

1. Secondary hypertension;
2. Severe hypertension or other antihypertensive drugs unable to be discontinued;
3. History of heart failure or record of LVEF < 40%, cardiomyopathy or valvular heart disease;
4. Severe arrhythmia, including arrhythmia, atrial fibrillation, atrial flutter, ventricular tachycardia, advanced atrioventricular block and sick sinus syndrome;
5. History of myocardial infarction or unstable angina during the past three months;
6. Type I diabetes;
7. Type II diabetes, fasting blood-glucose ≥ 11.1mmol/L;
8. ALT or AST ≥ 1.5 times the upper limit of the reference value;
9. Abnormal thyroid function (hyperthyroidism and hypothyroidism);
10. Acute or chronic renal insufficiency (serum creatinine of male patient > 176.8 μmol/L and female patient > 159.12μmol/L);
11. Patient suffers from anxiety or depression;
12. Mental disease or senile dementia;
13. Hypersensitivity to calcium channel blockers;
14. Pregnancy, lactation; women of child-bearing age use hormonal contraception, or perimenopause women receive hormone treatment;
15. History of drug or alcohol abuse within two years prior to enrollment;
16. Concomitant administration of the following CYP3A4 strong inhibitors: ketoconazole, itraconazole, nefazodone, triacetyloleandomycin, clarithromycin, ritonavir, nelfinavir. Or other CYP3A4 inhibitors: erythromycin, verapamil, saquinavir, fluconazole; inducers of drugmetabolizing enzymes of liver (phenytoin, carbamazepine, rifampicin and barbiturates);
17. Patient has suffered from cerebrovascular accident, severe trauma or undergone major operation;
18. BMI ≥ 30 kg/m2;
19. Participation in other clinical trials during the past three months;
20. Investigator judged the patient unsuitable to participate in this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 281 (Actual)
Dates: Start 2011-12; Primary Completion 2013-03 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in mean seated diastolic blood pressure in clinical after 6 weeks of treatment | 6 weeks
  after 6 weeks of treatment, the Changes from baseline in mean seated diastolic blood pressure in clinical will be compared between study drug and control drug

SECONDARY OUTCOMES:
Change from baseline in mean seated systolic blood pressure after 6 weeks of treatment | 6 weeks
  1. Change from baseline in mean seated systolic blood pressure after 6 weeks of treatment;
  2. Normalization rate
     * Normalization rate of clinical: defined as patients with a SBP<140mmHg and a DBP<90mmHg after 6 weeks of treatment.
     * Normalization rate of ABPM: defined as patients with mean BP < 130/80 mm Hg within 24 hours after 6 weeks of treatment.
     * Normalization rate of self-measurement: defined as patients with mean BP < 135/85 mm Hg within 1 week after 6 weeks of treatment.
  3. Analysis the heteromorphosis of BP and HR.
  4. Evaluate the total effective rate of clinical

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai First People's Hospital, Shanghai, China

REFERENCES:
- [Derived] Xu M, Wu Y, Wang H, Xu X, Zhao S, Zhang M, Jin H, Yan J, Wang B, Gong J, Lu X, Peng J, Dai Q. Effects of lercanidipine hydrochloride versus felodipine sustained-release on day-to-day home blood pressure variability. Curr Med Res Opin. 2016 Oct;32(sup2):43-52. doi: 10.1080/03007995.2016.1220932. PMID 27779454